CLINICAL TRIAL: NCT05408741
Title: A Pilot Study Assessing the Effectiveness of Use of Guided Imagery for Treatment of Pain and Symptom Management in Women With Post-mastectomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1104; NCI-2022-04827 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-05

CONDITIONS: Pain Syndrome; Pain; Symptom Management
MeSH Terms: conditions — Somatoform Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (The Intervention Group) (Experimental): Participants will receive guided imagery and deep breathing technique exercises.
  Interventions: Other: The Intervention Group
- Group 2 ( The Control Group) (Experimental): Participants will not receive any relaxation techniques. Participants will receive the current standard of care.
  Interventions: Other: The Control Group

INTERVENTIONS:
Other: The Intervention Group — Participants will complete a 20-minute guided imagery exercise (which includes deep breathing exercises) every day at home using the selected app and/or resource you downloaded at the beginning of this study.
  Arms: Group 1 (The Intervention Group)
Other: The Control Group — Participants will continue to receive your current care, but will not receive guided imagery or deep breathing exercises from a social worker.
  Arms: Group 2 ( The Control Group)

SUMMARY:
To learn if using guided imagery and deep breathing techniques can help with pain management in patients who have post-mastectomy pain syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objective:

-To evaluate the effectiveness of use of Guided imagery and deep breathing techniques in pain management compared to control arm in patients with post-mastectomy pain syndrome who don't receive intervention and only receive standard care.

Secondary objective:

To evaluate effectiveness of Guided imagery and deep breathing techniques in symptom cluster management including fatigue, sleep, depression, and anxiety and in general quality of life compared to control arm who don't receive intervention and only receive standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Breast Cancer patients who were performed mastectomy in previous 12 months
2. Post-mastectomy pain syndrome >4 weeks.
3. Patients who report 2-10 on the baseline pain severity score or 2-10 on the baseline pain interference score
4. Patients ≥ 18 years old and ≤ 70 years old
5. Must understand and read English, sign a written informed consent, and follow protocol requirements
6. If on medication for anxiety or depression, stable dose of medications for management of anxiety or depression symptoms for at least six weeks prior to enrollment with no plans to change medications in the subsequent four weeks. Increases or decreases allowed within drug class, but changing drug class will make patient in-evaluable

Exclusion Criteria:

1. Pending surgery during treatment
2. Suicidal ideation
3. Diagnosis of a formal thought disorder (e.g., schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
The change in pain severity score and the change in pain interference score, measured by brief pain inventory short form. Brief Pain Inventory: 0-10 No Pain-0 Worst Pain-10 | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Uzondu Osuagwu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT05408741/ICF_000.pdf